CLINICAL TRIAL: NCT05759585
Title: Examining the Effects of Person-centered Lifestyle Intervention in Individuals With Rheumatoid Arthritis: a Randomized Controlled Trial
Brief Title: Examining the Efficacy of Personalized Lifestyle Intervention in Individuals With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SULTAN BASTURK, professional, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-SBASTURK-001
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centered lifestyle intervention group (Experimental): Intervention group: Volunteers who were diagnosed with RA by a rheumatologist according to the 2010 criteria of the American College of Rheumatology (ACR)/European Rheumatology Association (ACR/EULAR) will be included in the study.
  Person-centered lifestyle intervention in individuals with rheumatoid arthritis is planned as 2 sessions per week, for a total of 4 weeks.
  Interventions: Behavioral: person-centered lifestyle intervention
- Control group (Experimental): Control group: Volunteers who were diagnosed with RA by a rheumatologist according to the 2010 criteria of the American College of Rheumatology (ACR)/European Rheumatology Association (ACR/EULAR) will be included in the study.
  For the control group, they will be called twice a week for 4 weeks and inquired about their general condition.
  Interventions: Behavioral: person-centered lifestyle intervention

INTERVENTIONS:
Behavioral: person-centered lifestyle intervention — Lifestyle intervention is a combined approach that encourages individuals to change their lifestyles by increasing participation in meaningful readings. This program aims to facilitate the individual's self-development of healthy routines and habits; It includes techniques such as patient education, occupational self-analysis, problem-solving, motivation generation, and implementation of behaviors to prevent and manage disease-related symptoms.

SUMMARY:
It is aimed to examine the effects of person-centered lifestyle intervention on occupational performance, general health status, and quality of life in individuals with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is defined as a chronic, inflammatory autoimmune disease that can damage both joints and non-articular organs, including the heart, kidneys, lungs, digestive system, eyes, skin, and nervous system.

Management of RA requires a multidisciplinary approach, as common risk factors for RA include both modifiable lifestyle-related variables and non-modifiable traits such as genetics and gender. Although there is no definitive cure, it is necessary to optimize physical, emotional, and social health in order to minimize the impact of the disease. At this point, self-management interventions come to the fore.

Since many areas of life are affected in individuals with RA, it is seen that there is a need for combined treatments that address the individual holistically, as suggested by EULAR. Lifestyle intervention is a combined approach that encourages individuals to change their lifestyles by increasing participation in meaningful readings. There is strong evidence in the literature that Lifestyle intervention is an effective approach to managing the symptoms of many chronic diseases.

The number of studies involving lifestyle interventions in individuals with RA, whose importance is emphasized in the literature, is limited. Therefore, our study was planned to examine the effects of person-centered lifestyle intervention on occupational performance, general health status, and quality of life in individuals with RA. Hypotheses:

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with RA between the ages of 18-65 and meeting the ACR/EULAR diagnostic criteria
* Patients with low to moderate disease activity (DAS28 ≤5.1)
* No pharmacological treatment changes for RA in the last 3 months
* Have not had any surgery in the last 6 months
* Understand and cooperate with testing guidelines
* to be literate

Exclusion Criteria:

* Having any musculoskeletal disease, neurological disease, and/or visual and auditory impairment other than RA
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measurement | change from baseline score at the end of 4 weeks and 6 months
  COPM is a standardized measurement tool that reflects the change in an individual's personal perception of activity performance and satisfaction over a period of time. It is designed to identify the activity performance problems of the individual, to give priority to these areas and to develop person-centered practice. In this assessment scale, activity performance problems faced by the person in the areas of self-care, productivity, play-free time are recorded with a semi-structured interview method. Among these areas, the person is asked to select 5 problems that he prioritizes and to rate each problem area between 1 and 10 points. A higher score on this rating indicates greater performance and satisfaction. The calculation is made by dividing the total performance and satisfaction score by the number of selected activities.

SECONDARY OUTCOMES:
The DAS 28 Disease Activity scale | change from baseline score at the end of 4 weeks and 6 months
  Disease Activity Score (DAS-28), which includes 28 joints, is used to monitor objective and subjective measures of disease activity in individuals with RA [33, 34]. The DAS-28 has been shown to have good validity and internal consistency reliability for monitoring this patient population [35] and is able to distinguish between patients with high and low disease activity [33]. Objective measures for rheumatoid arthritis are the number of swollen joints and the level of inflammation (erythrocyte sedimentation rate or C-reactive protein); subjective measures are the number of tender joints and the patient's overall health assessment. Disease activity scores range from 0 (not completely active) to 9.4 (very active). It is classified as ≤ 3.2 = mild, >3.2 to ≤5.1 = moderate, and >5.1 = severe [36].
Health Assessment Questionnaire (HAQ) | change from baseline score at the end of 4 weeks and 6 months
  Evaluate how an individual's health status affects their physical function. It consists of eight subsections containing 20 activities (dressing and preparation, sitting-standing, eating, walking, hygiene, reaching, grip strength, and other activities) and each subsection contains two or three questions. All questions are rated on a four-point likert (0=I can do it easily), and (3=I can't do it at all). Eight subdivision scores are added up and divided by eight. A high score indicates poor health [37]. The Turkish validity and reliability of the test was established [38].
Hospital Anxiety and Depression Scale (HADS) | change from baseline score at the end of 4 weeks and 6 months
  The hospital anxiety and depression scale was developed by Zigmond and Snaith in 1983 [39]. In our country, the validity and reliability study was carried out by Aydemir[15] in 1997 [40]. The scale is used to determine the risk of anxiety and depression in the patient, to measure its level and change in severity.
General Self-Efficacy Scale | change from baseline score at the end of 4 weeks and 6 months
  The General Self-Efficacy Scale - Turkish form is a valid and reliable tool for measuring the general self-efficacy of people aged 18 years and older who are at least primary school graduates. The scale consists of 17 items and a 5-point likert structure. Bandura argues that the perception of self-efficacy is one of the main determinants of human behavior and behavioral changes [43]. The use of the concept of self-efficacy in the formation and change of patients' health-related behaviors seems to be beneficial in the field of health. The Turkish validity and reliability study of the scale was carried out by Yıldırım and İlhan in 2010 [44].
Rheumatoid Arthritis Quality of Life Scale | change from baseline score at the end of 4 weeks and 6 months
  It is a disease-specific scale developed for patients with Rheumatoid arthritis and evaluates the quality of life multi-dimensionally. It consists of 30 questions prepared to be answered as yes/no. Scores range from 0 to 30, and high scores indicate poor quality of life [45]. The Turkish version of the RAQoL was used in this study [46].
The Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire (BRAF-MDQ) | change from baseline score at the end of 4 weeks and 6 months
  It was developed to evaluate the effect of fatigue in different dimensions in RA patients. In the questionnaire, 4 questions (questions 1-4) evaluate physical fatigue, 7 questions evaluate fatigue in activities of daily living (ADL), 5 questions evaluate cognitive fatigue (questions 12-16), and 4 evaluate emotional fatigue. There are 20 questions in total (questions 17-20). All questions except the first 3 questions are asked to be answered according to the 4-point Likert system (none, a little, a lot, and a lot). The questionnaire completed by the patient evaluates the last seven days. The patient can leave a total of 3 questions blank. But it should answer questions 1 and 2. The patient scores between 0-70. A high score indicates high fatigue [41]. A Turkish validity and reliability study was conducted [42].

CONTACTS AND LOCATIONS:
Overall Officials: TIMUR PIRILDAR, PROF, Study Director — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University Hafsa Sultan Hospital, Manisa, Turkey (Türkiye)